CLINICAL TRIAL: NCT00869726
Title: A Double-Blind, Placebo Controlled Multicentre Study To Evaluate The Efficacy And Safety Of MBP8298 In Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: A Study for Patients With Secondary Progressive Multiple Sclerosis
Acronym: MAESTRO-01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: BioMS Technology Corp. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12788; I3E-BM-MSAB (Other: Eli Lilly and Company); MBP8298-01 (Other: BioMS Technology Corp.)
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — MBP-8298

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dirucotide (Experimental)
  Interventions: Drug: dirucotide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dirucotide — 500mg, intravenous, dosed once every six months for 18 months
  Other Names: MBP8298; LY2820671
  Arms: Dirucotide
Drug: Placebo — intravenous, once every six months for 18 months
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether MBP8298 is effective and safe in the treatment secondary progressive multiple sclerosis.

Dirucotide is generic name for MBP8298.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of SPMS
* Absence of relapse in the 3mos prior to baseline
* EDSS of 3.5 - 6.5
* Pyramidal or Cerebellar FSS greater than or equal to 3
* A cohort of 100 HLA DR2/4 negative patients is required. Once enrollment to this cohort is complete, all further patients are required to be HLA DR2/4 positive.
* Informed consent
* Subject reliability and compliance

Exclusion Criteria:

* Diagnosis of Primary Progressive MS
* Subjects have previously received MBP8298
* Recent history of malignancy, with the exclusion on basal cell carcinoma.
* Steroid therapy within 30 days prior to first study specific procedure or any other treatment known to be used for putative or experimental MS treatment
* Therapy with beta-interferon, glatiramer acetate within 3 mos or mitoxantrone, cyclophosphamide, methotrexate, azathioprine, or any other immuno-modulating or immunosuppressive drugs including recombinant or non-recombinant cytokines or plasma exchange within 6 mos prior to performance of the first study-specific test, with the exception of corticosteroids or ACTH for relapse treatment.
* Initiation or discontinuation of therapy with 4-AP or 3,4-DAP at any time during the study period.
* History of anaphylactic/anaphlactoid reactions to glatiramer acetate
* Abnormal lab values at the Screening Visit deemed by the Investigator to be clinically significant
* Known allergy to Gadolinium-DTPA
* Treatment at any time with Cladribine, total lymphoid irradiation, monoclonal antibody treatment
* Treatment at any time wtih an altered peptide ligand
* Any conditions that could interfere with the performance of study specific procedures e.g.MRI
* Previous randomization to this study
* Known positivity for HIV, Hepatitis B, or Hepatitis C
* Participation in any other non-MS clinical trial within 30 days prior to performance of the first study specific test or any investigational therapy in the past 6 mos.
* Females who are breast feeding, pregnant or not using a medically approved method of contraception regularly
* Known or suspected current or past alcohol or drug abuse (within the last year)
* Any medical, psychiatric or other condition that could result in a subject not being able to give fully informed consent, or to comply with the protocol requirements
* Any other condition that, in the investigator's opinion, makes the subject unsuitable for participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2004-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Increase in the time to worsening of disability by Kurtzke Expended Disability Status (EDSS). | baseline, 3mos, 6mos, 9mos, 12mos, 15mos,18mos, 21mos, 24mos

SECONDARY OUTCOMES:
degree of change in EDSS | baseline, 24mos
Brain Atrophy by MRI | baseline, 12mos, 24mos
Activity analysis of T2 and Gadolinium enhancing lesions | 12mos and 24mos
Lesion burden | 12mos and 24mos
Degree of change in MS Functional Composite Index (MSFC) | baseline, 3mos, 6mos, 9mos, 12mos, 15mos, 18mos, 21mos, 24mos
Relapse rates | baseline, 3mos, 6mos, 9mos, 12mos, 15mos,18mos, 21mos, 24mos
Quality of life as measured by Short Form 36 (SF-36) or MSQoL54 | baseline, 6mos, 12mos, 18mos, 24mos

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon-Fri 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- St. Michaels Hospital, Toronto, Ontario, Canada
- Copenhagen University Hospital, Copenhagen, Denmark
- West Tallinn Central Hospital, Tallinn, Estonia
- Terveystalo Turku Kuvantaminen, Turku, Finland
- Heinrich Heine Universitaets, Düsseldorf, Germany
- Vecmilgravis Hospital, Riga, Latvia
- Maaslandziekenhuis, Sittard, Netherlands
- Hospital Duran I Reynals, Barcelona, Spain
- Karolinska Universitetssjukhus, Stockholm, Sweden
- Walton Hospital, Liverpool, United Kingdom